CLINICAL TRIAL: NCT01056445
Title: Hemodynamic Instability Following Carotid Artery Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Javad Kojuri, Shiraz Univ ersity of medical Sciences
Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 88-1239
Record Dates: First submitted 2010-01-19; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2008-03

CONDITIONS: Carotid Stenting
Keywords: Carotid artery stenting; Hemodynamic Instability; Valsalva Ratio
MeSH Terms: interventions — Valsalva Maneuver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carotid stenting and hemodynamic instability (Active Comparator): 27 patients undergone carotid stenting
  Interventions: Procedure: valsalva maneuver
- carotid stenting without hemodynamic instability (Active Comparator): no hemodynamic instability after carotid stenting
  Interventions: Procedure: valsalva maneuver

INTERVENTIONS:
Procedure: valsalva maneuver — valsalva maneuver after carotid stenting
  Arms: carotid stenting and hemodynamic instability
Procedure: valsalva maneuver — valsalva maneuver after carotid stenting
  Arms: carotid stenting without hemodynamic instability

SUMMARY:
Hemodynamic instability was controlled in 27 patient during carotid stenting and it was showed that hemodynamic instability can be predicted by Valsalva maneuver before stenting and hemodynamic instability have no prognostic effect on result of carotid stenting.

DETAILED DESCRIPTION:
One of the important complications of Carotid Artery Stenting (CAS) is post procedural hypotension and bradycardia referred to as Hemodynamic Instability (HI). However its incidence and contribution to short-term prognosis of patients have been of a large debate. In this study we aim to assess the incidence and predictive factors of HI and its role in mortality and morbidity of patients in short-term follow-up.

Materials and Methods: 27 patients were selected based on NASCET criteria and underwent CAS between September 2008 and September 2009. Continuous EKG monitoring & supine blood pressure (BP) was obtained before and after stent deployment and on the following day to detect HI defined as systolic BP≤90mmHg or heart rate≤60 beats per minute. Patients were asked to perform Valsalva maneuver before and after stent deployment. Valsalva ratio along with other demographic and procedural data was documented and compared between patients with and without incidence of HI.

Results: 17 patients (63%) developed HI after CAS. The degree of stenosis was found to have a significant correlation with occurrence of HI with P value<0.006. No other risk factor or demographic data showed any correlation with HI. Valsalva Ratio (VR) were significantly lower in HI group compared with non-HI group indicating a significant autonomic dysfunction (P<0.003). In the follow-up one (4.3%) patient had developed major stroke and others were symptom free.

Conclusion: HI occurs frequently following CAS but seems to be a benign phenomenon and doesn't increase the risk of mortality or morbidity after the procedure in short-term. VR at rest (VR≤1.10) baseline autonomic dysfunction and degree of carotid artery stenosis can be used as measures for prediction of HI after CAS.

ELIGIBILITY:
Inclusion Criteria:

* every patient with carotid stenting

Exclusion Criteria:

* presence of hemodynamic instability and low BP at baseline
* atrial fibrillation
* unstable patients with recent TIA and CVA in last week
* inability of patient to hold respiration for 30 seconds
* refusal of patient

Ages: 49 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
predictors of hemodynamic instability | 0, 1, 6 months

SECONDARY OUTCOMES:
result of carotid stenting | 0, 1, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: javad kojuri, M.D., Principal Investigator — shiraz University of medical asciences
Locations (1):
- Shiraz University of Medical Sciences, Cardiovascular Research Center, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Kojuri J, Ostovan MA, Zamiri N, Farshchizarabi S, Varavipoor B. Hemodynamic instability following carotid artery stenting. Neurosurg Focus. 2011 Jun;30(6):E12. doi: 10.3171/2010.12.FOCUS10219. PMID 21631213